CLINICAL TRIAL: NCT06875830
Title: Comparison of Flapless Immediate Implant Placement With Titanium Mesh Versus Immediate Implants Placement With Collagen Membrane in Type II Socket: A Randomized Clinical Trial
Brief Title: Comparison of Immediate Implant Placement With Titanium Mesh Versus Collagen Membrane in Type II Socket:
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Misr International University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: PER5253015
Record Dates: First submitted 2025-03-09; First posted 2025-03-13 (Actual); Last update posted 2026-01-13 (Actual); Status verified 2025-03

CONDITIONS: Bone Augmentation; Badly Broken Maxillary Premolars Indicated for Extraction

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- immediate implant with collagen membrane (Active Comparator): immediate implant placement will be done and augmentation of the buccal bone will be done with xenograft and collagen membrane
  Interventions: Procedure: collagen membrane
- immediate implant with titanium mesh (Active Comparator): immediate implant placement will be done and augmentation of the buccal bone will be done with xenograft and titanium mesh
  Interventions: Procedure: titanium mesh

INTERVENTIONS:
Procedure: collagen membrane — augmentation of the buccal plate of bone with xenograft and collagen membrane
  Arms: immediate implant with collagen membrane
Procedure: titanium mesh — augmentation of the buccal plate of bone with xenograft and titanium mesh
  Arms: immediate implant with titanium mesh

SUMMARY:
Statement of the problem: Immediate implant placement is faced with several problems. One of the most important issues is dealing with defects in the buccal plate of bone in the esthetic zone.

Aim: The aim of this study is to assess the buccal bone thickness after augmentation with titanium mesh and xenograft upon flapless immediate implant placement.

DETAILED DESCRIPTION:
Statement of the problem: Immediate implant placement is faced with several problems. One of the most important issues is dealing with defects in the buccal plate of bone in the esthetic zone.

Aim: The aim of this study is to assess the buccal bone thickness after augmentation with titanium mesh and xenograft upon flapless immediate implant placement.

Materials and Methods: This parallel arm, randomized controlled clinical trial will involve systemically free patients with remaining roots or badly decayed teeth in the anterior region and buccal bone deficiency requiring implant placement. They will be randomly allocated to two equal groups. Group A (test group, n=10) will receive immediate implants (grafting with xenograft covered by titanium mesh covered by collagen membrane), while group B (test group, n=10) will receive immediate implants (grafting with xenograft covered by collagen membrane). The parameters ( buccal bone thickness & soft tissue thickness will be assessed at 6 & 12 months. Postoperative pain and swelling will be recorded daily by the patient for the 1st two weeks post surgically. Postoperative medication will be prescribed to the patient and postoperative instructions will be explained in detail. Follow-up will be performed to assess the parameters and to ensure performing proper oral hygiene. Data collected will be tabulated and statistically analyzed.

ELIGIBILITY:
Inclusion Criteria:

1. Patients who have at least one remaining root or badly decayed tooth in anterior maxilla.
2. Systemically free patients (American Society of Anesthesiologists I; ASA I)
3. Patients aged from 21 to 50 years old
4. Buccal bone partial deficiency (extraction socket type II)
5. Good oral hygiene
6. Accepts the follow-up period (cooperative patients)
7. Patient accepts to provides an informed consent

Exclusion Criteria:

1. Patients with habits that may jeopardize the implant longevity and affect the results of the study such as parafunctional habits such as bruxism
2. Smokers
3. Pregnant and lactating females

Ages: 21 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 20 (Estimated)
Dates: Start 2025-03-06 (Actual); Primary Completion 2026-07-01 (Estimated); Study Completion 2026-09-01 (Estimated)

PRIMARY OUTCOMES:
Buccal bone thickness | at baseline, 6 and 12 months
  assessment of the Buccal bone thickness in mm using CBCT

SECONDARY OUTCOMES:
Soft tissue thickness | at baseline 6 and 12 months
  Soft tissue thickness will be assessed in mm using volumetric analysis method
Keratinized tissue width | at baseline, 6 and 12 months
  measurement of the keratinized tissue width in mm using periodontal probe

CONTACTS AND LOCATIONS:
Overall Officials: ahmed H Farid, Masters, Principal Investigator — Assistant lecturer
Locations (1):
- Faculty of oral & dental Medicine,Misr international University, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: No